CLINICAL TRIAL: NCT05892640
Title: Effects of Low Salt Dietary Intake on Th17-Mediated Inflammation and Vascular Reactivity in Patients With Psoriasis
Brief Title: Low-Salt Diet Effect on Th17-Mediated Inflammation and Vascular Reactivity in Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Ines Drenjancevic, Vice Dean for Science, Faculty of Medicine Josip Juraj Strossmayer University of Osijek, Josip Juraj Strossmayer University of Osijek
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 215861462341
Record Dates: First submitted 2023-05-27; First posted 2023-06-07 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Psoriasis Vulgaris
Keywords: Diet, Sodium-Restricted; Psoriasis; Laser-Doppler Flowmetry; Microcirculation; Endothelium
MeSH Terms: conditions — Psoriasis | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-Salt Diet (Experimental): Low-salt diet (LS diet) according to DASH eating plan, with sodium intake of 1500 mg (3.75 g of salt), within the period of 14 days
  Interventions: Other: Low-Salt Diet

INTERVENTIONS:
Other: Low-Salt Diet — Low-salt diet (LS diet) according to DASH eating plan, with sodium intake of 1500 mg (3.75 g of salt), within the period of 14 days

SUMMARY:
Psoriasis presents an independent cardiovascular risk factor characterized by chronic low-grade systemic inflammation and oxidative stress which altogether might lead to endothelial dysfunction. It has been reported that increased oxidative stress has a pivotal role in high dietary sodium-induced endothelial dysfunction. Previous studies on sodium accumulation in psoriatic skin lesions and the sodium-induced augmentation in Th17 immune response, raise the question on the complex interplay between sodium and psoriasis, especially in the context of cardiovascular morbidity.

This study aimed to investigate the effect of a 2-week low-salt diet on endothelium-dependent and endothelium-independent cutaneous microvascular vasodilation and Th17-Mediated Inflammation in patients with psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosed psoriasis vulgaris
* subjects do not use topical corticosteroid therapy for at least 2 weeks before inclusion in the study and 2 weeks during the study
* subjects do not use systemic or biological therapy for at least 3 months before and 2 weeks during the study.

Exclusion Criteria:

* age < 18 years
* existence of other immune-mediated diseases (with the exception of autoimmune thyroid diseases and psoriatic arthritis - people with these comorbidities can be included)
* malignant diseases
* current infectious diseases and allergic reactions within 6 weeks before the start of the study

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Microvascular endothelial function | 2 weeks
  Cutaneous microvascular blood flow will be measured by Laser Doppler Flowmetry in response to vascular occlusion (post occlusive reactive hyperaemia - PORH), in response to iontophoresis of acetylcholine (ACh) and local thermal hyperemia (LTH) before and after LS diet protocol
Frequency of peripheral T helper 17 (Th17) and regulatory lymphocytes (Treg) among parent lymphocytes sub-population | 2 weeks
  Flow cytometry assessment of the frequencies of peripheral Treg and Th17 lymphocytes before and after LS diet protocol

SECONDARY OUTCOMES:
Microvascular non-endothelial function | 2 weeks
  Cutaneous microvascular blood flow will be measured by Laser Doppler Flowmetry in response to iontophoresis of sodium nitroprusside (SNP) before and after LS diet protocol
Relative amount of serum- and glucocorticoid-induced kinase 1 (SGK1) in peripheral blood mononuclear cells | 2 weeks
  Relative amount of total serum- and glucocorticoid regulated kinase 1 (SGK1) in cultured cells will be measured by commercially available cell-based enzyme-linked immuno-sorbent assay (ELISA) kit before and after LS diet protocol
Serum Protein Concentration of Pro- and Anti-Inflammatory Cytokines | 2 weeks
  Serum protein concentrations (pg/mL) of pro-inflammatory and anti-inflammatory cytokines will be measured with panel for multiplex protein quantitation before and after LS diet protocol
24-hour natriuresis | 2 weeks
  A 24-h urinary sodium excretion will be measured in each participant before and after LS diet protocol in order to assess compliance to the given dietary protocol

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No